CLINICAL TRIAL: NCT02275169
Title: Follicle-stimulating Hormone Treatment for Infertile Male Patients With Non-obstructive Azoospermia: a Multicenter Randomized Clinical Trial
Brief Title: FSH Treatment for Non-obstructive Azoospermic Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Sanitaria Locale Bari (Other)
Collaborators: Minia University (Other)
Responsible Party: Principal Investigator, Ettore Caroppo, Dr, Azienda Sanitaria Locale Bari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASLBari
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Azoospermia
Keywords: follicle stimulating hormone treatment; azoospermia nonobstructive; male infertility; follicle stimulating hormone
MeSH Terms: conditions — Azoospermia; Azoospermia, Nonobstructive; Infertility, Male | interventions — Urofollitropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated (Experimental): Urofollitropin 150 IU ampoules three times a week for three months
  Interventions: Drug: Urofollitropin
- Controls (Placebo Comparator): Placebo ampoules three times a week for three months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Urofollitropin — Urofollitropin 75 IU 2 ampoules three times a week for three months
  Other Names: Fostimon
  Arms: Treated
Other: Placebo — Placebo ampoules administered three times a week for three months
  Arms: Controls

SUMMARY:
Aim of the study is to evaluate the effect of highly purified human follicle-stimulating hormone treatment on the chance of retrieving testicular sperm (sperm retrieval rate) from infertile male patients with non-obstructive azoospermia of unknown origin.

DETAILED DESCRIPTION:
Preliminary reports showed that hormonal treatment may improve the chance of retrieving viable testicular sperm from men with NOA, but no RCT are available in the field. This randomized placebo-controlled clinical trial sought to evaluate whether the testicular sperm retrieval rate could result higher in NOA patients treated with follicle-stimulating hormone compared to placebo-treated NOA subjects.

ELIGIBILITY:
Inclusion Criteria:

* Azoospermia;
* testis longitudinal axis less than 4.5 cm;
* serum follicle-stimulating hormone greater than 7.6 IU/L

Exclusion Criteria:

* History of testicular biopsy,
* malignancy,
* varicocele,
* hyperprolactinemia,
* thyroid disfunction,
* chemotherapy,
* radiotherapy

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Sperm retrieval rate (SRR) | three months
  testicular sperm retrieval rate after three months of urofollitropin treatment

SECONDARY OUTCOMES:
IVF pregnancy rate | three to six months
IVF implantation rate | three to six months

CONTACTS AND LOCATIONS:
Overall Officials: Ettore Caroppo, MD, Study Director — ASL Bari; Craig Niederberger, MD, Study Chair — University at Illinois at Chicago UIC College of Medicine; Alayman Hussein, MD, Principal Investigator — El Minia University

REFERENCES:
- [Background] Sussman EM, Chudnovsky A, Niederberger CS. Hormonal evaluation of the infertile male: has it evolved? Urol Clin North Am. 2008 May;35(2):147-55, vii. doi: 10.1016/j.ucl.2008.01.010. PMID 18423236
- [Background] Schoor RA, Elhanbly S, Niederberger CS, Ross LS. The role of testicular biopsy in the modern management of male infertility. J Urol. 2002 Jan;167(1):197-200. PMID 11743304
- [Result] Caroppo E, Niederberger C, Vizziello GM, D'Amato G. Recombinant human follicle-stimulating hormone as a pretreatment for idiopathic oligoasthenoteratozoospermic patients undergoing intracytoplasmic sperm injection. Fertil Steril. 2003 Dec;80(6):1398-403. doi: 10.1016/s0015-0282(03)02202-7. PMID 14667875
- [Result] Kato Y, Shiraishi K, Matsuyama H. Expression of testicular androgen receptor in non-obstructive azoospermia and its change after hormonal therapy. Andrology. 2014 Sep;2(5):734-40. doi: 10.1111/j.2047-2927.2014.00240.x. Epub 2014 Jun 12. PMID 24919724
- [Result] Hussein A, Ozgok Y, Ross L, Rao P, Niederberger C. Optimization of spermatogenesis-regulating hormones in patients with non-obstructive azoospermia and its impact on sperm retrieval: a multicentre study. BJU Int. 2013 Mar;111(3 Pt B):E110-4. doi: 10.1111/j.1464-410X.2012.11485.x. Epub 2012 Sep 7. PMID 22958644